CLINICAL TRIAL: NCT04689763
Title: The Effectiveness of Lifestyle Redesign Training in Elderly With Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201912EM017
Record Dates: First submitted 2020-12-29; First posted 2020-12-30 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Aging
Keywords: life-style activities; cognitive functions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle Redesign Training (Experimental): The participants will receive a total of 12 training sessions, and each session will contain 120 minutes of training.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training — The programs contain sequential cognitive and exercise training, health lectures, and groups of daily living participation. We plan to assess the participants before and after the intervention programs. We expect that elders receiving training will improve on outcome measures. The results of the study will provide evidence of interventions for elderly with cognitive decline.

SUMMARY:
Taiwan is already an aging society due to the rapid increase of the aging population. To cope with this situation, it is necessary to make preparations for the care of the elderly. World Health Organization (WHO) proposed aging health strategy in recent years, and the community participation is the most important for the elderly. The courses provided by the community empowering are important to promote the healthy life of the elderly. However, at this stage, there are relatively few courses related to cognitive functions, life-style activities and aging education. It is needed to add more courses related to multi-domain.

DETAILED DESCRIPTION:
Taiwan is already an aging society due to the rapid increase of the aging population. To cope with this situation, it is necessary to make preparations for the care of the elderly. World Health Organization (WHO) proposed aging health strategy in recent years, and the community participation is the most important for the elderly. The courses provided by the community empowering are important to promote the healthy life of the elderly. However, at this stage, there are relatively few courses related to cognitive functions, life-style activities and aging education. It is needed to add more courses related to multi-domain.

Investigators anticipate recruiting a total of 50 participants with cognitive decline. The participants will receive a total of 12 training sessions, and each session will contain 120 minutes of training. The programs contain sequential cognitive and exercise training, health lectures, and groups of daily living participation. Investigators plan to assess the participants before and after the intervention programs. Investigators expect that elders receiving training will improve on outcome measures. The results of the study will provide evidence of interventions for elderly with cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* able to follow instruction (MMSE>= 20)
* self- or informant-reported memory or cognitive complaint.

Exclusion Criteria:

* recent myocardial infarction,heart failure,recent heart surgery,
* severe asthma, concomitant with other neurological disorders, or joint deformity that might prevents them performing exercise or cognitive training.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change scores of the Montreal Cognitive Assessment (MoCA) | baseline, posttest (around 12 weeks after baseline)
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Change scores of Mini-Mental State Exam (MMSE) | baseline, posttest (around 12 weeks after baseline)
  The Mini-Mental State Examination (MMSE) is the most commonly administered psychometric screening assessment of cognitive functioning. The MMSE is used to screen patients for cognitive impairment, track changes in cognitive functioning over time, and often to assess the effects of therapeutic agents on cognitive function. The total score of MMSE ranged from 0 to 30. Higher values represent a better cognitive functioning.
Change scores of the Stroop test | baseline, posttest (around 12 weeks after baseline)
  The Stroop test will be used to assess the processing speed, inhibition, set-shifting, and selective attention abilities. The participants will be tested under 2 conditions: congruent and incongruent conditions. In the congruent condition, the color ink of a word is consistent with the written color name; while the color ink differs from the written color name under the incongruent condition.
Change scores of the Timed up and go (TUG) test | baseline, posttest (around 12 weeks after baseline)
  The TUG test will be used to assess the mobility and dynamic balance ability. The participants will be required to stand up from a chair, walk 3 meters, turn around, then walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers and frail elderly (Podsiadlo & Richardson, 1991). The test-retest reliability of TUG on individuals with cognitive impairment was excellent.
Change scores of the Dual-task test | baseline, posttest (around 12 weeks after baseline)
  The dual-task tests will be assessed to determine the ability for an individual to perform 2 tasks simultaneously. The investigators will assess the dual-task performance during walking and performing box and block test. The results of the dual-task tests will provide information regarding to whether the 2 tasks compete for the same class of neural resources or one of the tasks can be carried out automatically
Change scores of the Wechsler Adult Intelligence Scale (WAIS) | baseline, posttest (around 12 weeks after baseline)
  The dual-task tests will be assessed to determine the ability for an individual to perform 2 tasks simultaneously. The investigators will assess the dual-task performance during walking and performing box and block test. The results of the dual-task tests will provide information regarding to whether the 2 tasks compete for the same class of neural resources or one of the tasks can be carried out automatically
Change scores of the Lawton Instrumental Activities of Daily Living Scale (IADL) | baseline, posttest (around 12 weeks after baseline)
  Assess activities of daily living. There are 8 domains of function measured with the Lawton IADL scale, including ability to use phone,shopping, food preparation, housekeeping, laundering, mode of transportation, responsibility for own medications,and ability to handle finances. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent). For each category, circle the item description that most closely resembles the client's highest functional level (either 0 or 1).

SECONDARY OUTCOMES:
Change scores of the Community Integration Questionnaire (CIQ) | baseline, posttest (around 12 weeks after baseline)
  The social participation level will be assessed with the Community Integration Questionnaire (CIQ).It contains 15 items to evaluate the degree of integration into each of the three area of family, social network, and productive activities. The total scores range from 0 to 29 with larger numbers indicating better integration.
Change scores of Geriatric Depression Scale (GDS) | baseline, posttest (around 12 weeks after baseline)
  The Geriatric Depression Scale (GDS) - 15 items version is a self-administered questionnaire used to evaluate mood and depressive symptoms. The scores range is 0-15 and a score of 5 or greater taken as a possible indicator of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan